CLINICAL TRIAL: NCT03121118
Title: Return of Amyloid Imaging Results
Brief Title: Return of Amyloid Imaging Results (RAISR Study)
Acronym: RAISR
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer H. Lingler, Associate Professor, University of Pittsburgh
Other Study IDs: PRO13100338
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Amyvid; Amyloid Imaging; PET Brain Scan; Amyloid Plaque; Ethics; Results disclosure
MeSH Terms: conditions — Cognitive Dysfunction; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Scan opportunity: 40 dyads comprised of individuals with Mild Cognitive Impairment and a study partner who is either a family member or kin-like friend.
  Interventions: Other: Scan Opportunity
- Comparison group: 40 dyads comprised of individuals with Mild Cognitive Impairment and a study partner who is either a family member or kin-like friend.

INTERVENTIONS:
Other: Scan Opportunity — Participants in the scan group are provided the option of having an amyloid PET brain scan and receiving their results which can inform them of risk for developing Alzheimer's Disease.
  Groups: Scan opportunity

SUMMARY:
Diagnostic tests designed to detect Alzheimer's disease (AD) pathology are increasingly popular in research on cognitive aging and AD. Due to concerns that information from such tests may be misunderstood, psychologically harmful, and of unclear clinical significance, results of pre mortem tests of AD pathology have typically been withheld from research participants. However, as the reliability and potential clinical significance of tests like brain amyloid imaging have become clear, there is a pressing need to revisit the practice of unilaterally withholding such information from research participants and identify responsible approaches to communicating individual results. Amyloid imaging results may be particularly relevant to mild cognitive impairment (MCI), a population for whom a growing body of evidence suggests that such testing may provide valuable prognostic and planning information, despite the unavailability of interventions to alter one's clinical course. Our preliminary work suggests that research participants with MCI and their family members are receptive to and capable of understanding information about the purpose, results, and implications of amyloid imaging when presented using a standardized approach developed by our interdisciplinary team. Building on this work, the proposed study will examine a well characterized sample of MCI care dyads (patient + family member) who will be randomized to either receive the opportunity to decide if they would like to pursue an amyloid PET Scan, or be randomized to not receive that opportunity (and will serve in the no-scan comparison group). This study aims to test hypotheses that examine how receiving amyloid imaging results will impact understanding of, and perceived self-efficacy for coping with, MCI among both patients and care partners.

DETAILED DESCRIPTION:
Objective:

Advances in amyloid imaging are leading to unprecedented changes in research on cognitive aging. We intend to characterize the way individuals respond to learning of the results of their amyloid imaging scans, understand the context in which decisions to obtain results of brain amyloid status are made, and examine the impact of such knowledge over the first year following results disclosure.

Specific Aim:

To determine the effect of receiving amyloid imaging results on understanding of, and perceived efficacy to cope with, Mild Cognitive Impairment (MCI) as a potential precursor to dementia.

Hypothesis 1. MCI care dyads who receive amyloid imaging results, using the text and visual aids developed by our interdisciplinary team, will a) perform better on objective assessments of basic knowledge about MCI and its relation to AD, and b) report lower levels of perceived ambiguity about what MCI means, as compared to control MCI care dyads not receiving amyloid imaging.

Hypothesis 2. MCI care dyads who receive the patient's amyloid imaging results, using the text and visual aids developed by our interdisciplinary team, will report higher levels of perceived efficacy to cope with MCI as compared to those not participating in amyloid imaging.

Background: Amyloid imaging is a brain scanning technique that uses radioligands along with positron emission tomography (PET) to detect the presence of neuritic plaques associated with Alzheimer's disease (AD). Evidence accumulating over the past decade suggests that current imaging techniques show fibrillar amyloid beta deposits in patients with known AD in a pattern consistent with post mortem pathological descriptions of amyloid plaque distribution (1,2). Although the prognostic utility of amyloid imaging in cognitively healthy older adults remains unclear, it is increasingly evident that brain amyloid positivity may have significant implications for the long-term outcomes of individuals with mild cognitive impairment (MCI).

Across 5 published studies, 155 persons with both amnestic and other subtypes of MCI have received amyloid PET scans and been followed longitudinally (3-7). Of these 155 individuals, 101 were amyloid positive at baseline, just over half (n = 53) of whom converted to dementia within 1 to 3 years. By contrast, only 7.4% (n = 4) of those who were amyloid negative at baseline converted to dementia within the same time period.

This body of research suggests that, regardless of MCI subtype, amyloid imaging is a unique and powerful indicator of clinical outcomes in MCI. This mounting evidence of the prognostic value of amyloid imaging underscores the significance of providing amyloid research participants who have MCI with information about, and the choice of, receiving their amyloid PET scan results. It is recognized that such results are not medically actionable because there are no FDA-approved treatments for MCI or otherwise effective means of slowing progression to dementia.

Despite the fact that amyloid PET research results are not medically actionable in MCI, preliminary findings from our team's investigation of disclosing mock amyloid scan results to MCI care dyads (patient + family member) indicate that these individuals are highly receptive to and generally capable of understanding information about amyloid-based biomarkers for AD, including the limitations and limited clinical utility of such testing.

Significance: Amyloid imaging advances are leading to unprecedented changes in research on cognitive aging and AD. As the field transitions into an era of pre-mortem testing for AD pathology, amyloid imaging is playing a key role in identifying candidates for and evaluating effectiveness in anti-amyloid clinical trials. Whereas tests of cognitive function have long been the gold standard for measuring treatment response, amyloid-based markers are rapidly being adopted as secondary outcome measures and, in some cases, methodologies of choice for evaluating the effectiveness of experimental therapies targeting AD. In clinical practice, the recent FDA approval of the commercial amyloid imaging agent, florbetapir, suggests that in the near future tests of pre-mortem AD pathology, while not sufficient to render a dementia diagnosis, may augment clinical evaluations of cognitive impairment. Findings from this research will lead to guidelines to assist clinicians in counseling and supporting individuals who are considering undergoing such testing.

ELIGIBILITY:
Inclusion Criteria:

All MCI participants:

1. Participant at the Pittsburgh Alzheimer's Disease Research Center, or other cognitive impairment studies.
2. Carry a current diagnosis of MCI
3. Have a family member or kin-like friend who also signs informed consent to participate
4. Female participants must be 5 years post menopausal by self-report

All family member participants:

1) At least 18 years of age 2) Can read and write English

-

Exclusion Criteria:

All MCI patient participants:

1. familial AD genetic mutation carriers (this group already has biomarker-derived knowledge of their dementia risk)
2. evidence of active, untreated primary psychiatric disorders defined as a CES-D (Depression Rating Scale) score of >=16 or a Spielberger State Anxiety score of >40 (to minimize the possibility of adverse events and to reduce any confounding influence of baseline mood)
3. Active suicidal ideation indicated via the Beck Scale for Suicidal Ideation and verified by clinician interview.

Participants with MCI and their primary participating family member:

1) Inability to provide direct consent to the study based on performance on the University of San Diego Brief Assessment of Capacity to Consent (meaning, proxy consent will not be accepted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 mild cognitive impairment dyads (patient + family member or kin-like friend). Mild cognitive impairment can consist of isolated impairment in memory; isolated deficit in non-memory domain; or, mild deficits in multiple cognitive domains.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Understanding of mild cognitive impairment as a potential precursor to dementia--knowledge | One month followup
  Score on a knowledge questionnaire
Understanding of mild cognitive impairment as a potential precursor to dementia-Coherence | One month followup
  Score on Brief Illness Perception Questionnaire Coherence Subscale
Perceived efficacy to cope with mild cognitive impairment as a potential precursor to dementia | One month followup
  Score on Coping Self-Efficacy Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Lingler, RN, PhD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim H, Lingler JH. Disclosure of amyloid PET scan results: A systematic review. Prog Mol Biol Transl Sci. 2019;165:401-414. doi: 10.1016/bs.pmbts.2019.05.002. Epub 2019 Jun 13. PMID 31481171
- [Background] Lingler JH, Butters MA, Gentry AL, Hu L, Hunsaker AE, Klunk WE, Mattos MK, Parker LS, Roberts JS, Schulz R. Development of a Standardized Approach to Disclosing Amyloid Imaging Research Results in Mild Cognitive Impairment. J Alzheimers Dis. 2016 Mar 8;52(1):17-24. doi: 10.3233/JAD-150985. PMID 27060950
- [Result] Lingler JH, Sereika SM, Butters MA, Cohen AD, Klunk WE, Knox ML, McDade E, Nadkarni NK, Roberts JS, Tamres LK, Lopez OL. A randomized controlled trial of amyloid positron emission tomography results disclosure in mild cognitive impairment. Alzheimers Dement. 2020 Sep;16(9):1330-1337. doi: 10.1002/alz.12129. Epub 2020 Jun 26. PMID 32588971
- [Result] Mattos MK, Sereika SM, Beach SR, Kim H, Klunk WE, Knox M, Nadkarni NK, Parker LS, Roberts JS, Schulz R, Tamres L, Lingler JH. Research Use of Ecological Momentary Assessment for Adverse Event Monitoring Following Amyloid-beta Results Disclosure. J Alzheimers Dis. 2019;71(4):1071-1079. doi: 10.3233/JAD-190091. PMID 31322563
- [Result] Lingler JH, Roberts JS, Kim H, Morris JL, Hu L, Mattos M, McDade E, Lopez OL. Amyloid positron emission tomography candidates may focus more on benefits than risks of results disclosure. Alzheimers Dement (Amst). 2018 May 30;10:413-420. doi: 10.1016/j.dadm.2018.05.003. eCollection 2018. PMID 30094328